CLINICAL TRIAL: NCT00989170
Title: Family Program for Weight Gain Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08-1206
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Program for the Prevention of Weight Gain (Experimental): Use of an enhanced Family Program on the prevention of weight gain in families with overweight children.
  Interventions: Behavioral: Family Program for the Prevention of Weight Gain
- No enhanced Family Program (Active Comparator)
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Family Program for the Prevention of Weight Gain — The Family Workbook is a step-by-step instruction guide for families to use throughout the 6-month period, detailing healthy lifestyle. All handouts, instructions, activities, and a timeline of the program are laid out for families in this workbook.
  Arms: Family Program for the Prevention of Weight Gain
Behavioral: Control Group — This group will not be provided the workbook and it is hypothesized those in the control group will gain excess weight.
  Arms: No enhanced Family Program

SUMMARY:
The long-term goal of this project is to develop, evaluate, and disseminate to Extension Service families across the state of Colorado, an engaging, interactive, and evidence-based Family Program in order to prevent weight gain in adults and excess weight gain in children. Excess weight gain in children is defined as an increase in body weight beyond the increase in weight associated with normal growth and development. The program will focus on small, easily adopted, sustainable, lifestyle changes.

Project Objectives include:

1. Enhancing a Family Program by including food and physical activity environmental assessments, an online social network, and a pre-programmed health-based text messaging system, and by gaining feedback from extension families through a series of 6 focus groups.
2. Conducting a randomized trial to evaluate the impact of the enhanced Family Program on the prevention of weight gain in families with overweight children. The investigators hypothesize that excess weight gain will be prevented in subjects in the intervention group, while those in the control group will gain excess weight.
3. Disseminating the Family Program through USDA Cooperative Extension Services in Colorado and evaluate the usefulness/effectiveness of the program for USDA Extension agents and participating families. The investigators will conduct 4 additional focus groups at the end of this objective to gain feedback on its usefulness in a "real-life" setting. This objective is different from objective 2 in that the investigators are evaluating the program in a real-life setting, using qualitative and self-reported data, rather than conducting a clinical trial.

By conducting focus groups with Extension families during both objectives #1 and 3, the Family Program will help to improve knowledge regarding behavioral and environmental factors influencing obesity. After enhancing the Family Program (Objective #1), the investigators will test its effectiveness in a randomized study of 200 families (Objective #2). Finally, after having developed and tested this effective intervention strategy, the investigators will disseminate it through Extension Agents throughout the state to evaluate its usefulness in a "real-life" setting (Objective #3).

ELIGIBILITY:
Inclusion Criteria:

* Families with at least one overweight child (8-12 years of age, BMI for age between the 84.6th and 95.4th percentile)

Exclusion Criteria:

* Individuals with physical or medical limitations that prevent them from engaging in physical activity. We will screen potential subjects and exclude subjects with an underlying disease that would inhibit activity using the Physical Activity Readiness Questionnaire (PAR-Q)
* Individuals using medication that influences body weight and appetite such as ADHD medication (e.g. Ritalin) and medication for depression.
* Pregnant and lactating women because their patterns of physical activity and eating may be different from their usual baseline. In the event a woman becomes pregnant during the study her data will not be included in the final analyses.
* Adults or children who are weight unstable due to weight loss surgery, weight loss medication, or dietary behavior.
* Families who do not have access to the internet at home or are not willing or able to use public access computers e.g., libraries and schools.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the randomized study is the proportion of overweight children who gain BMIp during the 6-month study period. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: James Hill, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Center for Human Nutrition, Denver, Colorado, United States